CLINICAL TRIAL: NCT03608488
Title: The Effect of Vitamin D and Exercise on Balance in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tugbaozsoy
Record Dates: First submitted 2018-07-04; First posted 2018-08-01 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency
Keywords: balance; vitamin D; exercise; fall risk
MeSH Terms: conditions — Vitamin D Deficiency; Motor Activity | interventions — Vitamin D; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D<10 ng/ml; Vitamin D replacement (Experimental): Vitamin D replacement (50.000 IU/per week, for 8 weeks)
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D<10 ng/ml; Vitamin D replacement and exercise (Experimental): Vitamin D replacement (50.000 IU/per week, for 8 weeks) and Core and balance exercises for 8 weeks.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D<10 ng/ml; exercise (Experimental): Core and balance exercises for 8 weeks.
  Interventions: Other: Exercise
- Vitamin D>30ng/ml; exercise (Active Comparator): Core and balance exercises for 8 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D3 50.000 IU/per week, for 8 weeks
  Other Names: exercise
  Arms: Vitamin D<10 ng/ml; Vitamin D replacement; Vitamin D<10 ng/ml; Vitamin D replacement and exercise
Other: Exercise — Core stability, balance exercises
  Arms: Vitamin D<10 ng/ml; exercise; Vitamin D>30ng/ml; exercise

SUMMARY:
In recent years, skeletal and nonskeletal effects of vitamin D has been studied. One of the effects of it was balance and fall prevention. However, these studies were performed on older patients who had not vitamin D deficiency. This study aimed to evaluate the effect of vitamin D replacement therapy and exercise on balance in 50-70 years-old postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 years-old postmenopausal women
* Vitamin D level<10 ng/ml and Vitamin D level>30 ng/ml
* Independant in daily life
* Able to do exercise
* Able to read and write in Turkish

Exclusion Criteria:

* Diabetes mellitus,
* Polyneuropathy,
* Spinal stenosis,
* History of fracture or lower extremity operation,
* Rheumatologic diseases,
* History of chemotherapy
* Cognitive impairment

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Ozsoy-Unubol, MD, Principal Investigator — Sultan Abdulhamid Han Training and Research Hospital
Locations (1):
- Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise: Vitamin D: Vitamin D3 50.000 IU/per week, for 8 weeks and Exercise: Core stability, balance exercises
Period: Overall Study
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Started | 22 | 21 | 22 | 45
Completed | 21 | 18 | 20 | 40
Not Completed | 1 | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise | Total
Number analyzed (Participants) | 21 | 18 | 20 | 40 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 4 | 7
  >=65 years | 20 | 17 | 19 | 36 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.76 (5.08) | 54.66 (5.59) | 55.70 (4.84) | 58.82 (5.84) | 56.78 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 20 | 40 | 99
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 21 | 18 | 20 | 40 | 99
Region of Enrollment [Number; unit: participants]
  Turkey | 21 | 18 | 20 | 40 | 99

OUTCOME MEASURES:

1. Primary Outcome: Postural Stability Test (Biodex) Assessed at Baseline
Description: overall stability index: quantifying the ability to maintain dynamic postural stability The patient's score on this test assesses deviations from center, thus lower index means less instability and better balance.
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.
  0 is the minimum score, but there is no defined maximum score
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score | 2.25 (1.27) | 2.30 (0.97) | 2.18 (1.01) | 1.97 (1.02)

2. Primary Outcome: Postural Stability Test (Biodex) Assessed After Treatment (8 Weeks)
Description: overall stability index: quantifying the ability to maintain dynamic postural stability.
  The patient's score on this test assesses deviations from center, thus a lower score is more desirable than a higher score.
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System 0 is the minimum score, but there is no defined maximum score
Time Frame: After treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score | 1.90 (1.20) | 1.83 (0.83) | 1.56 (0.74) | 1.43 (0.86)

3. Primary Outcome: Berg Balance Test Assessed at Baseline
Description: 14-item scale designed to measure balance of the older adult in a clinical setting minimum: 0 maximum: 56 A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score on a scale | 51.52 (2.94) | 51.77 (1.80) | 52.35 (1.59) | 53.02 (2.49)

4. Primary Outcome: Berg Balance Test Assessed After Treatment (8weeks)
Description: as for outcome 3
Time Frame: After treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score on a scale | 53.33 (2.67) | 53.55 (1.78) | 54.25 (1.37) | 54.27 (1.96)

5. Secondary Outcome: Fall Risk Assesment Performed at Baseline
Description: Biodex fall risk screening test: Patients were instructed to maintain the vertical projection with their center of gravity in the midpoint of the platform 0 is the best possible value, higher score reflects increased risk of falling. But there is no defined maximum score
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score | 1.69 (1.08) | 1.96 (0.94) | 1.90 (0.98) | 1.71 (0.98)

6. Secondary Outcome: Fall Risk Assesment Performed After Treatment (8 Weeks)
Description: Biodex fall risk screening test: Patients were instructed to maintain the vertical projection with their center of gravity in the midpoint of the platform 0° is the best possible value, higher score reflects increased risk of falling. But there is no defined maximum score.
Time Frame: After treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score | 1.40 (0.74) | 1.57 (0.69) | 1.35 (0.57) | 1.81 (2.79)

7. Secondary Outcome: Health Status Assessed at Baseline
Description: Notthingham Health Profile: general patient reported outcome measure which measures subjective health status.
  38 questions in 6 subareas, with each question assigned a weighted value; the sum of all weighted valuesin a given subarea adds up to 100. Overall score is calculated by summing up 6 subdomian scores.
  Ovearall minimum: 0 maximum: 600 (6X100) Higher scores reflect worse health status
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score on a scale | 263.35 (143.52) | 212.81 (137.78) | 229.98 (119.31) | 161.10 (109.88)

8. Secondary Outcome: Health Status Assessed After Treatment (8 Weeks)
Description: as for outcome 7
Time Frame: After treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
Number analyzed (Participants) | 21 | 18 | 20 | 40
score on a scale | 170.19 (120.24) | 158.23 (145.94) | 171.98 (108.18) | 119.30 (97.04)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed.
Arm/Group | Vitamin D<10 ng/ml; Vitamin D Replacement | Vitamin D<10 ng/ml; Exercise | Vitamin D<10 ng/ml; Vitamin D Replacement and Exercise | Vitamin D>30ng/ml; Exercise
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03608488/Prot_SAP_000.pdf